CLINICAL TRIAL: NCT02101203
Title: A Double-blind, Randomized, Placebo-controlled, Dose-finding Study to Investigate the Safety and Efficacy of Lybridos in the Domestic Setting in Healthy Female Subjects With Hypoactive Sexual Desire Disorder and Maladaptive Activity of Sexual Inhibitory Mechanisms
Brief Title: Lybridos in Pre-and Postmenopausal Women With Hypoactive Sexual Desire Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emotional Brain NY Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EB90a extension
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: HSDD
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Experimental): 40 subjects administered placebo
  Interventions: Drug: Placebo
- Testosterone + Buspirone (Experimental): 40 subjects administered 0.5 mg Testosterone + 10 mg Buspirone hydrochloride
  Interventions: Drug: 0.5 mgTestosterone + 10 mg Buspirone

INTERVENTIONS:
Drug: Placebo
  Other Names: Solid Oral Dosage. Maximum every other day (on an as needed basis)
  Arms: Placebo
Drug: 0.5 mgTestosterone + 10 mg Buspirone — A total of 28 doses will be provided. Subjects are required to take a minimum of 8 doses over the 8-week treatment period (1 dose/week). The other 20 doses may be taken as desired (ie, "on demand") throughout the 8-week treatment period; dosing is permitted every 2 days (ie, on alternate days).
  Other Names: Solid Oral Dosage. Maximum every other day (on an as needed basis)
  Arms: Testosterone + Buspirone

SUMMARY:
A double-blind, randomized, placebo-controlled, dose-finding study to investigate the safety and efficacy of Lybridos in the domestic setting in healthy female subjects with hypoactive sexual desire disorder and maladaptive activity of sexual inhibitory mechanisms.

This is a 2-arm placebo and Lybridos (0.5 mg testosterone + buspirone 10 mg) extension to study EB90 (Clinical Study Protocol EB90a, version 3.0, 07 June 2013).

In the present study, the efficacy of Lybridos will be evaluated in the domestic setting in healthy female subjects with HSDD and maladaptive activity of sexual inhibitory mechanism(s). Sexual satisfaction and other aspects of sexual functioning will be measured within 24 hours after each sexual activity. The following hypotheses will be tested:

Lybridos, as compared to placebo, will significantly increase the number of satisfying sexual events.

Objectives:

To investigate the efficacy of Lybridos as compared to placebo in increasing the number of satisfactory sexual episodes in healthy female subjects with hypoactive sexual desire disorder (HSDD) and maladaptive activity of sexual inhibitory mechanisms

* To identify the optimal dose of Lybridos to take into phase 3 clinical development
* To confirm that Lybridos has superior efficacy as compared to testosterone alone and to buspirone alone
* To evaluate the effect of Lybridos as measured by scales of sexual satisfaction and/or sexual desire/arousal
* To evaluate the safety profile of Lybridos

DETAILED DESCRIPTION:
None entered

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

1. Provision of written informed consent
2. Females between 21 and 70 years of age, inclusive, pre or postmenopausal, with HSDD (comorbidity with female sexual arousal disorder [FSAD] and/or female orgasmic disorder [FOD; only as secondary diagnosis] is allowed). The diagnosis of HSDD will be established by a trained health care professional.
3. Maladaptive activity of sexual inhibitory mechanism(s) (see appendix 4 for definition)
4. Be involved in a stable relationship and have a partner who will be at home for the majority of the study duration
5. Healthy according to normal results of medical history, physical examination, laboratory values, and vital signs; exceptions may be made if the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible to participate in the study:

Cardiovascular Conditions

1. Any underlying cardiovascular condition, including unstable angina pectoris, that would preclude sexual activity
2. Systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure > 90 mmHg. For subjects ≥ 60 years old and without diabetes mellitus, familial hypercholesterolemia, or cardiovascular disease: systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 90 mmHg
3. Systolic blood pressure ≤ 90 mmHg and/or diastolic blood pressure ≤ 50 mmHg Gynecological and Obstetric Conditions
4. Use of any contraceptive containing anti-androgens (e.g. Cyproteron acetate) or (anti)androgenic progestogens (drospirenone, dienogest, chlormadinone acetate and norgestrel)
5. Use of any contraceptive or hormone replacement therapy (HRT) containing more than 50 μg/day of estrogen
6. Positive test result for Chlamydia or gonorrhea
7. Pregnancy or intention to become pregnant during this study (Note: A urine pregnancy test will be performed in all women of child bearing potential prior to the administration of study medications.)
8. Lactating or delivery in the previous 6 months prior to signing Informed Consent Form
9. Significant abnormal Pap smear in the previous 12 months prior to signing Informed Consent Form
10. History of bilateral oophorectomy
11. Other unexplained gynecological complaints, such as clinically relevant abnormal uterine bleeding patterns
12. Perimenopausal status (cycle shortening/irregular menstrual bleeding in the last 12 consecutive months and/or occurrence of vasomotor symptoms (e.g. hot flashes, night sweating) in combination with elevated FSH levels (>40 IU/L) for women from age 40 onwards; in women with a history of hysterectomy perimenopausality can be assessed by FSH levels (>40 IU/L) and/or vasomotor symptoms Other Medical Conditions
13. Liver and/or renal insufficiency (aspartate aminotransferase, alanine aminotransferase and gamma glutamyltransferase > 3 times the upper limit of normal and/or estimated glomerular filtration rate (eGFR) < 60.00 mL/min based on the Cockcroft Gault formula)
14. Any current endocrine disease or endocrinopathy (e.g. uncontrolled thyroid dysfunction) as determined by medical history, basic physical examination and/or laboratory values significantly outside the normal range of the central laboratory; or uncontrolled diabetes mellitus(HbA1c > 7.5%)
15. Free- and/or total testosterone levels outside the upper limit of the reference range of the central laboratory (free testosterone: > 1.1 ng/dL, and total testosterone > 80 ng/dL)

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the number of satisfactory sexual episodes, measured using the Sexual Satisfaction of an Event Questionnaire (SSEQ). | 20 weeks
  Sexual satisfaction will be evaluated based on a global satisfaction assessment comparing the 4-week establishment period with the 8 week DB treatment period. In addition there is a 8 week run in period between the establishment period and the double blind treatment period for a total treatment period of 20 weeks.

SECONDARY OUTCOMES:
Sexual Satisfaction | 20 weeks
  Sexual satisfaction will be evaluated based on a global satisfaction assessment comparing the 4-week establishment period with the 8 week DB treatment period. In addition there is a 8 week run in period between the establishment period and the double blind treatment period for a total treatment period of 20 weeks
Sexual desire and arousal | 20 weeks
  Sexual desire and arousal will be evaluated based on the 'desire' and 'arousal' domains of the Sexual Anamnesis Questionnaire, the Sexual Function questionnaire and weekly diaries throughout the course of the study.
Sexual Distress | 20 weeks
  Sexual Distress will be assessed using the Female Sexual Distress Scale-Revised (FSDS-R).
Subjective evaluation of gain and improvement | 20 weeks
  Using the following tools, perceived gain and improvement will be assessed:
  * Subjective Evaluation of Gain (SEG)
  * Subjective Evaluation of Improvement (SEI)
  * Patient's Global Impression of Improvement (PGI-I)
  * Patient Benefit Evaluation (PBE)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - San Diego Sexual Medicine, San Diego, California
  - Meridien Research, Bradenton, Florida
  - Compass Research, Orlando, Florida
  - Meridien Research, St. Petersburg, Florida
  - Comprehensive Clinical Trials LLC, West Palm Beach, Florida
  - Annapolis Sexual Wellness Center, Annapolis, Maryland
  - Maryland Center for Sexual Wellness, Lutherville, Maryland
  - Maryland Primary Care Physicians, Queenstown, Maryland
  - NECCR Fall River LLC, Fall River, Massachusetts
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania